CLINICAL TRIAL: NCT02481700
Title: Epidemiological Study on the Surgical Removal of Third Molars
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S57824
Record Dates: First submitted 2015-06-22; First posted 2015-06-25 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Impacted Third Molar Tooth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Third molar removal — The surgical removal of third molars

SUMMARY:
The aim of this study is to get a clear view on current practice of surgical third molar removal in Belgium and the association with morbidity and complications.

For this prospective cohort study, patients who visit the outpatient department of Oral and Maxillofacial Surgery of the University Hospitals Leuven or hospitals affiliated with the Flemish Hospital Network will be participating. All included patients are referred from primary dental providers for the surgical removal of one or more third molars. Before participating, written informed consent will be recorded from all eligible subjects.

Patients consult one of the oral and maxillofacial surgeons or residents working on the department of the University Hospitals Leuven for the removal of third molars. In the standard procedure, patients are not routinely clinically monitored after one week at the department.

Pre-operative, operative and postoperative data will be collected through a questionnaire, extracted data from the patient's medical file and panoramic radiography. The surgeon's individual operation technique will be registered through a one-off questionnaire. The questionnaires are taken at the same time of consultation and includes a maximum of 8 questions per time and are considered as non-invasive and a minimal burden for the patient. Postoperatively, patients record their recovery status and ability to resume daily- and work activities at day 3 and 10 by using a dairy system and, if necessary, revisit the outpatient department of oral and maxillofacial surgery.

ELIGIBILITY:
Inclusion Criteria:

* referred for the removal of one or more third molars

Exclusion Criteria:

* other concomitant oral procedures in the same surgical session

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All included patients are referred from primary dental providers for the surgical removal of one or more third molars
Sampling Method: Probability Sample
Enrollment: 6010 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Morbidity | 10 days
  Assessing pain, trismus, swelling and neurosensory disturbances

SECONDARY OUTCOMES:
Resuming daily activities | 10 days
  Household, work, studies